CLINICAL TRIAL: NCT01263964
Title: Troponin Elevation in Acute Ischemic Stroke (TRELAS) - a Prospective Study on the Frequency and Correlation to Coronary Artery Disease and to Stroke Localisation
Brief Title: Troponin Elevation in Acute Ischemic Stroke (TRELAS)
Acronym: TRELAS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christian Nolte, PD Dr.med., Charite University, Berlin, Germany
Other Study IDs: EA4/118/10; 01 EO 0801 (Other Grant/Funding Number: German Ministry of Research and Education)
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Stroke
Keywords: ischemic stroke; troponin elevation; transient apical ballooning; acute coronary syndrome; troponin elevation,; culprit lesion on coronary angiogram,; troponin elevation and stroke localisation (temporal lobe?)
MeSH Terms: conditions — Stroke; Ischemic Stroke; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers indicating myocardial or neuronal damage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- stroke, troponin elevation: Patients with stroke (proven by cerebral imaging) and troponin elevation undergoing coronary angiogram
  Interventions: Procedure: coronary angiogram
- non-stemi (controll group): Patients with troponin elevation suggesting non-stemi undergoing coronary angiogram
  Interventions: Procedure: coronary angiogram

INTERVENTIONS:
Procedure: coronary angiogram — coronary angiogram

SUMMARY:
The primary objective of the prospective observational trial TRELAS (TRoponin ELevation in Acute ischemic Stroke) is to elucidate the underlying pathomechanism of cTnT elevation in acute ischemic stroke. Consecutive patients with acute ischemic stroke admitted to the Department of Neurology Campus Benjamin Franklin of the university hospital Charité will be screened for cTnT elevations suggestive of myocardial infarction (>0,05 µg/l). Patients with increased troponin will undergo diagnostic coronary angiography within 72 hours. Diagnostic findings of coronary angiographies taken out in age- and gender-matched patients presenting with NSTE-ACS (Non-ST-Elevation Acute Coronary Syndrome) to the Division of Cardiology will serve as a control. The primary endpoint of the study will be the occurrence of culprit lesions indicating focal cardiac damage on the basis of an acute CAD.

DETAILED DESCRIPTION:
The primary objective of the prospective observational trial TRELAS (TRoponin ELevation in Acute ischemic Stroke) is to elucidate the underlying pathomechanism of cTnT elevation in acute ischemic stroke in order to give guidance for clinical practise. All consecutive patients with acute MRI- or CT-confirmed ischemic stroke admitting within 72 hours after symptom onset to the Department of Neurology Campus Benjamin Franklin of the university hospital of the Charité will be screened for cTnT elevations suggestive of myocardial infarction (>0,05 µg/l) on admission and day 2. Patients with increased troponin will undergo diagnostic coronary angiography within 72 hours. Diagnostic findings of coronary angiographies taken out in age- and gender-matched patients presenting with NSTE-ACS (Non-ST-Elevation Acute Coronary Syndrome) to the Division of Cardiology will serve as a control. The primary endpoint of the study will be the occurrence of angiographic culprit lesions indicating focal cardiac damage on the basis of an acute CAD. Secondary endpoints will be the localisation of stroke in the cerebral imaging and ventriculographic findings of wall motion abnormalities suggestive of neurally mediated global cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke, confirmed by cerebral MRI or CT, respectively
2. Inclusion within ≤ 72 hours after symptom onset
3. hsTroponin T >0,05 µg/l

Exclusion Criteria:

1. Renal insufficiency (creatinine ≥1,2 mg/dl)
2. Limited life expectancy or mRS ≥ 4 prior to stroke event leading to hospital admission
3. Contraindications for the coronary angiography
4. Age < 18 years
5. Pregnancy
6. Patient unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted because acute ischemic stroke and additional troponin-elevation(cases) or non-stemi (controlls)
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
culprit lesion on coronary angiogram | 24 months

SECONDARY OUTCOMES:
transient apical ballooning on levocardiogram | 24 months
stroke localization | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Endres, Professor, Study Director — Charite Universitätsmedizin-Berlin
Locations (2):
- Germany (2):
  - Charite Campus Benjamin Franklin, Berlin, Germany
  - Charite, Campus Benjamin Franklin, Berlin, State of Berlin

REFERENCES:
- [Derived] Mochmann HC, Scheitz JF, Petzold GC, Haeusler KG, Audebert HJ, Laufs U, Schneider C, Landmesser U, Werner N, Endres M, Witzenbichler B, Nolte CH; TRELAS Study Group. Coronary Angiographic Findings in Acute Ischemic Stroke Patients With Elevated Cardiac Troponin: The Troponin Elevation in Acute Ischemic Stroke (TRELAS) Study. Circulation. 2016 Mar 29;133(13):1264-71. doi: 10.1161/CIRCULATIONAHA.115.018547. Epub 2016 Mar 1. PMID 26933082
- [Derived] Scheitz JF, Mochmann HC, Nolte CH, Haeusler KG, Audebert HJ, Heuschmann PU, Laufs U, Witzenbichler B, Schultheiss HP, Endres M. Troponin elevation in acute ischemic stroke (TRELAS)--protocol of a prospective observational trial. BMC Neurol. 2011 Aug 8;11:98. doi: 10.1186/1471-2377-11-98. PMID 21824425